CLINICAL TRIAL: NCT06223555
Title: Variability In Mixed Meal Tests: Fixed Versus Adjusted to Energy Needs Caloric Dose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 10001707; 001707-DK
Record Dates: First submitted 2024-01-24; First posted 2024-01-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12-15

CONDITIONS: Obesity; Healthy Volunteer
Keywords: Healthy Volunteer; Obesity; Body Composition; Diet; Mixed Meal Test; Glucose
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Fixed Mixed Meal Test
  Interventions: Other: Fixed Mixed Meal Test
- 2 (Active Comparator): Adjusted Mixed Meal Test
  Interventions: Other: Adjusted Mixed Meal Test

INTERVENTIONS:
Other: Fixed Mixed Meal Test — a FIXED dose meal that will be 900 kcal of a liquid meal
  Arms: 1
Other: Adjusted Mixed Meal Test — a body weight ADJUSTED dose liquid meal.
  (30% of total daily energy requirements)
  Arms: 2

SUMMARY:
Background:

Researchers use mixed meal tolerance tests (MMTTs) to look at how people s bodies respond to eating a meal. However, researchers do not agree on how to decide the number of calories to give in each meal. Some use fixed meals, which are the same size for everyone, and some use adjusted meals, based on the size of the person s body. Researchers want to know which MMTT is best to use for future research.

Objective:

To learn how fixed vs adjusted meals affect blood glucose levels in healthy people.

Eligibility:

Healthy people aged 18 years or older.

Design:

Participants will have 3 or 4 clinic visits of up to 8 hours in 8 weeks.

Participants will have baseline tests:

Their height, weight, and waist size will be measured.

They will have an oral glucose tolerance test: A needle attached to a tube (IV) will be inserted into a vein in the arm. They will have a sugary drink. Blood samples will be taken from the tube at intervals up to 3 hours after the drink.

They will have a body scan.

Participants will have 2 MMTT visits. One will include a fixed meal and one will include an adjusted meal. They will have tests at both visits:

Resting metabolic rate: A clear hood will be placed over the participant s head while they rest for 20 minutes. This will measure the oxygen they breathe in and out.

MMTT. Participants will have 5 minutes to drink a liquid meal. Blood samples will be taken at intervals for the next 4 hours....

DETAILED DESCRIPTION:
Study Description:

This study will be an outpatient study completed in 3-4 separate visits. We will compare two methods of dosing (fixed and adjusted) a mixed meal tolerance test (MMTT) to determine which results in greater physiological variability in hormone response. Ultimately, the goal is to determine which method of dosing is more appropriate in a research setting.

Objectives:

Primary Objective:

To determine whether an adjusted energy dose MMTT or a fixed dosed meal will result in greater variability in glucose area under the curve (AUC) within the same participants across a range of BMIs.

Secondary Objectives:

To determine whether baseline body composition, blood parameters (lipids, hormones, etc), and resting metabolic rate are associated with MMTT responses and whether this association is moderated by MMTT condition (fixed vs. adjusted).

Endpoints:

Primary Endpoint: Glucose area under the curve (AUC)

Secondary Endpoints: Area under the curve (AUC), incremental area under the curve (iAUC), value and timing of the absolute maximum (peak), value and timing of the inflection point after the absolute maximum value, value and timing of the maximum rate of incline, value and timing of the maximum rate of decline, total number of critical points with body composition, blood parameters, and resting metabolic rate as predictors.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form.
* Agreement to adhere to Lifestyle Considerations throughout study duration.
* Males and females; Age >= 18years
* Healthy, as determined by medical history, physical examination, and laboratory tests.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

* Current use of medications, dietary supplements, or alternative therapies known to alter energy metabolism.
* Fasting plasma glucose >= 126 mg/dL
* Type I or Type II Diabetes Mellitus by self-report.
* Hematologic disorders including significant anemia (male hemoglobin < 13.0 g/dL or female hemoglobin < 11.0 g/dL)
* Current pregnancy, pregnancy within the past 6 months or currently lactating
* History or self-report of gastrointestinal disease, including inflammatory bowel diseases (e.g. Chron s disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active) which may alter metabolism or absorption of study food by self-report
* Evidence of alcohol abuse as defined by an 8-point score on the Alcohol consumption screening AUDIT questionnaire in adults.
* Participants who report taking large doses of acetaminophen (> 3 grams daily) who cannot stop acetaminophen 24 hours prior to and following the meal tests will be excluded from the study.
* Inability to consume provided food based on a food allergy or intolerance.
* Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators.
* Any disorder, unwillingness, or inability not covered by any other exclusion criteria which, in the investigator s and/or team s opinion, jeopardizes the safety of the participant or others or would interfere with adherence to the protocol (such as claustrophobia).

Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine whether an adjusted energy dose MMTTor a fixed dosed meal will result in greater variability in glucose area under the curve (AUC) within the same participants across a range of BMIs. | Baseline, Visit 3/4
  Glucose AUC associated with MMTT conditions (fixed vs. adjusted).

SECONDARY OUTCOMES:
Body Composition | Baseline, Visit 3/4
  Change in energy expenditure associated with MMTT conditions (fixed vs. adjusted).
Resting Metabolic Rate | Baseline, Visit 3/4
  Change in energy expenditure associated with MMTT conditions (fixed vs. adjusted).
Lipids | Baseline, Visit 3/4
  Change in energy expenditure associated with MMTT conditions (fixed vs. adjusted).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Votruba, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001707-DK.html